CLINICAL TRIAL: NCT06313099
Title: Examination of the Parameters Regarding The General Health Status of Prison Officers
Brief Title: Parameters of the General Health Status of Prison Officers
Status: Completed | Type: Observational
Sponsor: Pakize Nurgul Sen (Other)
Responsible Party: Sponsor-Investigator, Pakize Nurgul Sen, Research Assistant, Sakarya Applied Sciences University
Organization: Sakarya Applied Sciences University (Other)
Other Study IDs: SakaryaAppliedSciencesUPNSC
Record Dates: First submitted 2024-03-08; First posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Musculoskeletal Pain; Fatigue; Depression; Quality of Life
MeSH Terms: conditions — Musculoskeletal Pain; Fatigue; Depression | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All participants will be evaluated
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — Participants' musculoskeletal system disorders were assessed using the Cornell Musculoskeletal Disorders Questionnaire (CMDQ), fatigue levels were measured using the Fatigue Severity Scale (FSS), sleep quality was evaluated using the Visual Analog Scale (VAS), depression levels were assessed using the Beck Depression Inventory (BDI), and quality of life was measured with the Nottingham Health Profile (NHP). Google Forms was used to create the data collection tools, which were then sent to the participants' email addresses and collected online.

SUMMARY:
Introduction The working conditions of prison officers are very stressful. Today, it is known that stress affects the health status of individuals in many ways. In this study, it was aimed to evaluate the musculoskeletal system problems, fatigue severity, depression levels, and quality of life of prison officers and to examine the relationship between these parameters and the socio-demographic characteristics of the participants.

Method The study included a total of 141 volunteers. The musculoskeletal problems of the participants were evaluated with the Cornell Musculoskeletal Disorders Questionnaire, fatigue levels were evaluated with the Fatigue Severity Scale, depression levels were evaluated with the Beck Depression Inventory, and quality of life was evaluated with the Nottingham Health Profile.

DETAILED DESCRIPTION:
The working conditions of prison officers are very stressful. Today, it is known that stress affects the health status of individuals in many ways. In this study, it was aimed to evaluate the musculoskeletal system problems, fatigue severity, depression levels, and quality of life of prison officers and to examine the relationship between these parameters and the socio-demographic characteristics of the participants.The study included a total of 141 volunteers. The prison management allowed the collection of data online due to the COVID-19 pandemic.141 prison officers between the ages of 18 and 65, working in Mula E Type Closed Penitentiary Institution, having completed at least one year in the profession and volunteering to participate in the study, participated in the research. Individuals who had received physical therapy in the last three months, had undergone surgery for an orthopedic reason in the last year, and had used pain medication for the last 15 days were not included in the study. The musculoskeletal problems of the participants were evaluated with the Cornell Musculoskeletal Disorders Questionnaire, fatigue levels were evaluated with the Fatigue Severity Scale, depression levels were evaluated with the Beck Depression Inventory, and quality of life was evaluated with the Nottingham Health Profile.

The Cornell Musculoskeletal Disorders Questionnaire consists of Likert-type questions inquiring about the painful region, the severity of pain, and the level of impact on work life for an individual. A total of 12 regions, starting from the neck area to the foot area, are examined. Each body region is scored on a scale ranging from 0 to 90. The Fatigue Severity Scale consists of 9 questions, with the lowest score being 9 and the highest score being 63. If the average of the scores obtained from these 9 questions is above 4, it indicates pathological fatigue. Participants were asked to consider the time from going to bed to falling asleep, the frequency of waking up after falling asleep, and the total time spent asleep. The Beck Depression Inventory consists of 21 questions, each scored between 0 and 3. The scores obtained from the scale are categorized into four groups. In the classification of the severity of depression, up to 9 points are considered no depression, 10-16 points are considered mild, 17-29 points are considered moderate, and 30-63 points are considered severe depression. The cutoff score for depression is accepted as 17.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-65
* Working in Muğla E Type Closed Penitentiary Institution
* Having completed at least one year in the profession
* Volunteering to participate in the study participated in the research.

Exclusion Criteria:

* Had received physical therapy in the last three months
* Had undergone surgery for an orthopedic reason in the last 1 year
* Had taken painkillers for the previous fifteen days.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 141 volunteer officers, ranging in age from 18 to 65, who were employed at Muğla E Type Closed Prison were included in the study.
Sampling Method: Probability Sample
Enrollment: 141 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-02-15 (Actual); Study Completion 2021-03-02 (Actual)

PRIMARY OUTCOMES:
Cornell Musculoskeletal Disorders Questionnaire | Through study completion, an average of 2 mounths
  Cornell Musculoskeletal Disorders Questionnaire: The questionnaire consists of Likert-type questions inquiring about the painful region, severity of pain and the level of impact on work life for an individual. A total of 12 regions, starting from the neck area to the foot area, are examined. Each body region is scored on a scale ranging from 0 to 90. The higher the score obtained from the questionnaire, the more significant the individual's musculoskeletal problems are presumed to be

SECONDARY OUTCOMES:
Fatigue Severity Scale | Through study completion, an average of 2 mounths
  Fatigue Severity Scale (FSS): The scale consists of 9 items, with the minimum score being 9 and the maximum score being 63. A higher score indicates a higher severity of fatigue. If the average score derived from these 9 items is above 4, it signifies the presence of pathological fatigue.
Sleep Quality: Virtual Analog Scala: VAS | Through study completion, an average of 2 mounths
  A Visual Analog Scale (VAS) was utilized to assess participants' sleep quality. Participants were asked to consider the time it took to fall asleep, the frequency of awakenings after falling asleep, and the total duration of sleep. A score of 0 indicated very poor sleep quality, while 10 indicated very good sleep quality.
Beck Depression Inventory | Through study completion, an average of 2 mounths
  The Beck Depression Inventory consists of 21 items, each scored between 0 and 3. As the score increases, the individual's level of depression rises. Scores obtained from the inventory are categorized into four groups. For the classification of depression severity, scores up to 9 indicate no depression, scores between 10 and 16 indicate mild depression, scores between 17 and 29 indicate moderate depression, and scores between 30 and 63 indicate severe depression. The cutoff score for depression is considered to be 17.
Nottingham Health Profile | Through study completion, an average of 2 mounths
  The scale consists of a total of 6 sections: physical activity, pain, sleep, social isolation, emotional reaction and energy level, comprising a total of 38 questions. Each section is scored between 0 and 100. Total score ranges from 0 to 600. A lower total score indicates a higher quality of life, while a higher total score suggests a poorer quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Muğla E Type Closed Prison, Muğla, Menteşe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No